CLINICAL TRIAL: NCT01022320
Title: Effect of Lateral Pharyngoplasty on Blood Pressure in Obstructive Sleep Apnea Patients
Brief Title: Effect of Lateral Pharyngoplasty on Blood Pressure in Obstructive Sleep Apnea (OSA) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Carolina Ferraz de Paula Soares, HSPE
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0024.0.338.000-09; HSPE-001/09 (Registry Identifier: Otorhinolaryngology department of HSPE)
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Obstructive Sleep Apnea; High Blood Pressure
Keywords: OSA; Blood pressure; Lateral Pharyngoplasty
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical outcome (Experimental): 20 consecutive cases of patients who underwent the lateral pharyngoplasty
  Interventions: Procedure: Lateral Pharyngoplasty

INTERVENTIONS:
Procedure: Lateral Pharyngoplasty — surgery lateral pharyngoplasty: consists on the section and rotation of the superior constrictor pharyngeal muscle associated with the ressection of the palatopharyngeus preserving the palatoglossus and mucosa of posterior and anterior tonsilar pillar , bilaterally.

SUMMARY:
* Describe blood pressure changes on patients with OSA treated with lateral pharyngoplasty
* Compare the mean of systolic and diastolic blood pressure in 24 hours, average systolic and diastolic pressure during daytime and night and changes in the nocturnal decrease.

DETAILED DESCRIPTION:
The variables are:

Ambulatory blood pressure data Snoring scale BMI neck circumference abdominal circumference medications and life style changes

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient
* BMI < 35
* no Benzodiazepinec User

Exclusion Criteria:

* BMI > 35
* Use of benzodiazepinecs
* Clinical contra-indications to surgery (ASA III or ASA IV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Soares, MD, Principal Investigator — HSPE
Locations (1):
- Hospital do Servidor Estadual de São Paulo, São Paulo, São Paulo, Brazil